CLINICAL TRIAL: NCT06023901
Title: The Importance of Mechanosensitive Cell Mediated Prostaglandin and Nitric Oxide Synthesis in the Pathogenesis of Apical Periodontitis: Comparative with Chronic Periodontitis
Brief Title: The Importance of Prostaglandin and Nitric Oxide Synthesis in Apical Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Seyda Ersahan, DDS, PhD, Principal Investigator, Clinical Associate Professor, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: E-10840098-772.02-2860/344
Record Dates: First submitted 2023-08-29; First posted 2023-09-05 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2023-08

CONDITIONS: Periapical Periodontitis
Keywords: Gingival crevicular fluid; Apical periodontitis; Chronic periodontitis
MeSH Terms: conditions — Periapical Periodontitis; Chronic Periodontitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 85 patients with only apical periodontitis (AP group) (Experimental): AP group was divided into 3 subgroups. AS-PAI 1 (mild): those having at least 1 tooth with either PAI 3 or PAI 4, AS-PAI 2 (moderate): those having only 1 tooth with a PAI 5, AS-PAI 3 (severe): those having two or more teeth with a PAI 5.
  Interventions: Diagnostic Test: Apical periodontitis
- 50 patients with only chronic periodontitis (CP group), (Experimental): In this study, the CP group was divided into 4 subgroups according to the periodontitis staging system (PSS) (Tonetti). This system classifies the periodontitis from I to IV according to the interdental clinical attachment loss (CAL), radiographic bone loss (RBL) and tooth loss. This scoring is as follows: Stage 1: CAL 1 to 2 mm, RBL is at coronal third (<15%) and no tooth loss, Stage 2: CAL 3 to 4 mm, RBL is at coronal third (15% to 33%) and no tooth loss, Stage 3: CAL > 5 mm, RBL is extending to mid-third of root and beyond and tooth loss < 4 teeth, and Stage 4: CAL > 5 mm, RBL is extending to mid-third of root and beyond and tooth loss > 5 teeth. However, Stage 1 and 2 were evaluated in the same group due to the low number of cases. As a result, the groups were designed as Stage 1-2: PSS 1-2, Stage 2: PSS 2 and Stage 3: PSS 3.
  Interventions: Diagnostic Test: Apical periodontitis
- A healthy control group of 50 volunteers (No Intervention): control group. A healthy control group of 50 volunteers without periodontal pathology as well as any acute/chronic disease (muscle/joint/bone diseases, inflammatory bowel disease, local or generalized infection, severe organ disease, cardiovascular disease and diabetes mellitus) were included in the study.

INTERVENTIONS:
Diagnostic Test: Apical periodontitis — Radiography of the patients were taken. Blood samples were collected from those patient
  Other Names: Chronic periodontitis
  Arms: 50 patients with only chronic periodontitis (CP group),; 85 patients with only apical periodontitis (AP group)

SUMMARY:
A total of 185 subjects were divided into three categories: AP group (n=85), CP group (n=50) and healthy control group (n=50). The AP group was divided into 3 subgroups according to abscess scoring (AS-PAI) based on the periapical index. The CP group was divided into 4 subgroups according to the periodontitis staging system (PSS). After recording the demographic and clinical characteristics of all participants, blood and gingival crevicular fluid (GCF) samples were taken. TNF-α, IL-10, PGE2 and NO levels were measured in these samples.

DETAILED DESCRIPTION:
* Study Design This observational, analytical, cross-sectional study was conducted at a single center. In order to reach the planned sample size, approximately 1200 patients who applied to the Department of Endodontics of xxxx university between June 2021 and May 2022 due to apical periodontitis (AP) and/or chronic periodontitis (CP) were recorded including their intraoral examination and demographic characteristics. As a result of the examination, 85 patients with only AP (AP group) and 50 patients with only CP (CP group), whose diagnosis was confirmed, were included in the study. Patients having both AP and P were excluded from the study. Patients who had taken antibiotics and/or anti-inflammatory drugs within the last 6 months and those with pregnancy or lactation were also excluded. In addition, those with a history of using steroid or nonsteroidal anti-inflammatory drugs and high-dose biotin vitamin in the last 48 hours were excluded from the study, as this may affect the results. A healthy control group of 50 volunteers without periodontal pathology as well as any acute/chronic disease (muscle/joint/bone diseases, inflammatory bowel disease, local or generalized infection, severe organ disease, cardiovascular disease and diabetes mellitus) were included in the study. Those included in the research groups; randomly selected from people with similar gender, age and weight characteristics.
* Demographic-Clinical History Gender, age, body mass index (BMI), comorbidity status of all patients participating in the study were recorded. The patients' root canal treatment (RCT), dental crown, composite/amalgam fillings (CF), number of missing teeth (NMT) findings were obtained as a result of intraoral examination.
* Periapical and Periodontal Disease Scoring All teeth present in the oral cavity were radiographed and the presence of radiolucent images associated with the periapical region and radiographic bone loss was assessed. Panoramic radiographs, in the study, were obtained using a digital panoramic unit (VistaPano S, Durr Dental AG, Germany), operating at 73kVp and 10 mA with 13500 milliseconds exposure time in standard mode. For periapical radiographs Carestream RVG 5200 (RVG; Carestream Health Inc, Atlanta, CA, USA) system was used with an x-ray unit, setting of 70 kV, 8 mA. The bisecting angle technique was applied in obtaining the periapical images. Then, the radiographs were analyzed with Kodak Dental Imaging Software. From radiographic evaluation of the teeth, the presence of periapical radiolucency without periodontal disease was considered sufficient for AP diagnosis. Abscess scoring (AS-PAI) based on the periapical index was performed as an indicator of disease progression within the AP group. For this scoring, the periapical index (PAI) scoring system,10 which is a scoring system for the radiographic evaluation of apical periodontitis, was used. Accordingly, the AP group was divided into 3 subgroups. AS-PAI 1 (mild): those having at least 1 tooth with either PAI 3 or PAI 4, AS-PAI 2 (moderate): those having only 1 tooth with a PAI 5, AS-PAI 3 (severe): those having two or more teeth with a PAI 5.

Periodontal measurements, obtained for the study, consisted of the highest probing depths (in milimetres) recorded around six selected teeth per participant. In this study, the CP group was divided into 4 subgroups according to the periodontitis staging system (PSS) (Tonetti). This system classifies the periodontitis from I to IV according to the interdental clinical attachment loss (CAL), radiographic bone loss (RBL) and tooth loss. This scoring is as follows: Stage 1: CAL 1 to 2 mm, RBL is at coronal third (<15%) and no tooth loss, Stage 2: CAL 3 to 4 mm, RBL is at coronal third (15% to 33%) and no tooth loss, Stage 3: CAL > 5 mm, RBL is extending to mid-third of root and beyond and tooth loss < 4 teeth, and Stage 4: CAL > 5 mm, RBL is extending to mid-third of root and beyond and tooth loss > 5 teeth. However, Stage 1 and 2 were evaluated in the same group due to the low number of cases. As a result, the groups were designed as Stage 1-2: PSS 1-2, Stage 2: PSS 2 and Stage 3: PSS 3.

• Collection of Venous Blood and Gingival Crevicular Fluid (GCF) Fasting (8-10 hours) venous blood of all participants was taken from forearm antecubital/basic veins. After keeping the blood at room temperature for 30 minutes, it was centrifuged at 2500 xg for 10 minutes. After centrifugation, the upper serum of the tubes was separated. Hemolysis indices (HI) of the sera were measured to prevent optical interference. (Cobas 8000 Chemistry Analyzer, USA). Those with a hemolysis index greater than 50 (mg/dl Hb) were excluded from the study. Appropriate sera were stored at -80oC until the day of analysis. In addition to venous blood, gingival crevicular fluid (GCF) samples were also collected and were stored at -80oC under similar conditions. On the day of analysis, all serums and GCF were first allowed to dissolve slowly at +4 oC and then brought to room temperature before measurement.

Gingival crevicular fluid samples were taken prior to periodontal probing to avoid contamination by blood. To avoid contamination of the sample, patients were asked not to eat or drink anything for at least 30 minutes before the procedure. Three samples were taken from the mesial, distal and buccal surfaces of related tooth. The selected sites were isolated with cotton roll and supragingival plaque, if present, was removed using a curette to prevent saliva and/or plaque contamination. GCF was collected for 60 seconds using PerioPaper strips (OraFlow Inc., NY, USA) placed gently until slight resistance was felt. The three samples were pooled into Eppendorf tubes and then placed in the laboratory freezer at -80 °C for storage. Periopapers were thoroughly washed in 0.5 ml eppendorf Tubes (after subtracting the tare weight of the tube) with 100 µl of phosphate-buffered saline (PBS) using an automatic pipette. Blood-stained paper strips were removed from the samples. All GCF samples were weighed on a precision balance (Shimadzu Libror, Model AEG-220, Germany) and recorded. All samples were thoroughly mixed with a 15-20 sec vortex device (Heidolph Reax Top Vortex, Schwabach, Germany). This allowed GCF to pass into PBS. The paper strips were removed without contaminating the samples and the remaining extract was stored in the freezer until the working day. The results obtained on the study day were proportioned by weights/PBS.

• Biochemical Analyzes TNF-α, IL-10, NO and PGE2 levels in the sera of all patients were measured in Microplate ELISA Reader (BioTek Epoch 2 Microplate ELISA Reader, USA) using the ELISA method. Due to the insufficient amount of sample (100 µl), only NO and PGE2 levels were measured in the GCF using the same ELISA kit.

Serum TNF-α, IL-10, NO and PGE2 levels were analyzed using ELISA plates whose wells were pre-coated with antibody (human TNF-α, IL-10, NO or PGE2). The sensitivity of TNF-α, IL-10, NO and PGE2 test kits (Bioassay Technology Laboratory, China) is 1.52 ng/L, 2.59 pg/mL, 1.12 µmol/L and 1.28 ng/L, measuring range 3-900 ng/L, respectively, 5-1500 pg/mL, 2-600 µmol/L and 2-600 ng/L, CV for all tests for intraassay and interassay were < 10%.

ELIGIBILITY:
Inclusion Criteria:

* Apical periodontitis (AP) and/or chronic periodontitis (CP)
* Patients who had taken antibiotics and/or anti-inflammatory drugs within the last 6 months - - Without periodontal pathology as well as any acute/chronic disease (muscle/joint/bone diseases, inflammatory bowel disease, local or generalized infection, severe organ disease, cardiovascular disease and diabetes mellitus) were included in the study

Exclusion Criteria:

* with pregnancy or lactation were also excluded.
* with a history of using steroid or nonsteroidal anti-inflammatory drugs and high-dose biotin vitamin in the last 48 hours were excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2022-01-02 (Actual); Study Completion 2023-08-02 (Actual)

PRIMARY OUTCOMES:
The inflammatory markers TNF-α, IL-1β, IL-6 and IL-10,17 | Through study completion, an average of 1 year
The biomarkers with protective functions such as PGE2 and NO2 | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Faculty of Dentistry, Istanbul, ESENLER, Turkey (Türkiye)